CLINICAL TRIAL: NCT05755542
Title: Occurrence of Long-Covid in Patients After Inpatient Rehabilitation Due to Acute Covid-19 Infection. How Easy is it for Patients to Return to Everyday Life and Work After Inpatient Rehabilitation Due to Acute Covid-19-infection?
Brief Title: Long-Covid in Patients Post Rehabilitation Treatment and Reintegration Into Everyday Life
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rehazentrum Walenstadtberg (Other)
Responsible Party: Sponsor
Other Study IDs: Covid Outcome
Record Dates: First submitted 2023-03-01; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the first study is to investigate how often a long Covid syndrome occurs after an inpatient rehabilitation due to previous hospitalization because of after acute Covid and whether there might be a connection with the severity during acute illness. 3 clusters of acute cases have been identified to be studied with regard to the long-term symptoms

1. Mild course (medication, oxygen)
2. Moderate course (IPS-IMC with NIV but without intubation)
3. Severe course (intubation)

The aim of the second study is to use a catamnestic survey and subsequent evaluation of the information to gain an insight into the existing functional deficits relevant to everyday life and restriction of the ability to participate in the workplace after rehabilitation treatment. The assessment of functional deficits is carried out in relation to:

1. Deficits in everyday skills (ADLs)
2. Restrictions in the ability to participate in the profession.

DETAILED DESCRIPTION:
All patients who had been infected with Walenstadtberg after acute Covid infection were included.

Patients were hospitalized for inpatient rehabilitation in the period from 01.04.2020 to 30.06.2022.

A written follow-up survey was carried out with regard to a possible persistent long Covid symptoms and possible persistent deficits in everyday skills and Restrictions in the ability to participate in the profession. There are 2 cohort studies.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* treated at a rehabilitation facility after being hospitilized for covid-19 infection
* complete questionnaire
* written consent to use collected data

Exclusion Criteria:

* < 18 years
* incomplete questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and Women over 18 years of age who have been treated at Rehazentrum Walenstadtberg after being hospitilized primarily because of an acute Covid-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-03-20 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Occurance of Symptoms pointing at Long-Covid after rehabilitation treatment | 2 years
  Occurance of Symptoms pointing at Long-Covid after rehabilitation treatment
Occurance of deficits in managing everyday life and work after covid infection | 2 years
  Investigation of deficits experienced by patients who have been treated at a rehabilitation facility after beeing hospitilized for a covid-19 infection and the impact of these deficits in everday life as well as in the workplace

SECONDARY OUTCOMES:
reinfection with covid-19 after rehabilition treatment | 2 years
  reinfection with covid-19 after rehabilition treatment
Impact of Covid-19 infection on quality of life | 2 years
  Impact of Covid-19 infection on quality of life in patients who have been treated at a rehabilition facility after beeing hospitilized due to a covid-19 infection

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Bachman, Prof., Study Director — Rehazentrum Walenstadtberg

IPD SHARING:
Plan to Share IPD: No